CLINICAL TRIAL: NCT00656747
Title: MAESTRAL - A Prospective, Multinational, Multicenter, Randomized, Double Blind, Double Dummy, Controlled Study Comparing the Efficacy and Safety of Moxifloxacin to That of Amoxicillin Clavulanic Acid for the Treatment of Subjects With Acute Exacerbations of Chronic Bronchitis.
Brief Title: Moxifloxacin Versus Amoxicillin Clavulanic Acid in Treatment of Acute Exacerbation of Chronic Bronchitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11980; 2007-006096-37 (EudraCT Number)
Record Dates: First submitted 2008-04-04; First posted 2008-04-11 (Estimated); Last update posted 2014-12-01 (Estimated); Status verified 2014-11

CONDITIONS: Chronic Bronchitis
Keywords: Chronic Obstructive Pulmonary Disease (COPD); Acute exacerbation of COPD (AECOPD); chronic bronchitis; bronchitis; chest infection; smoking; lung disease; lung; lungs
MeSH Terms: conditions — Bronchitis, Chronic; Pulmonary Disease, Chronic Obstructive; Bronchitis; Smoking; Lung Diseases | interventions — Moxifloxacin; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 2 (Active Comparator)
  Interventions: Drug: Amoxicillin clavulanic acid
- Arm 1 (Experimental)
  Interventions: Drug: Avelox (Moxifloxacin, BAY12-8039)

INTERVENTIONS:
Drug: Avelox (Moxifloxacin, BAY12-8039) — Subjects will be randomised to moxifloxacin 400 mg PO OD (5 days). Subjects will also take placebo tablets, so that each subject takes 3 tablets per day for 7 days. Prior to randomization, subjects are stratified based on co-administration of short-course systemic steroids.
  Arms: Arm 1
Drug: Amoxicillin clavulanic acid — Subjects will be randomised to amoxicillin-clavulanic acid 875/125 mg PO BID (7 days). Subjects will also take placebo tablets, so that each subject takes 3 tablets per day for 7 days. Prior to randomization, subjects are stratified based on co-administration of short-course systemic steroids.
  Arms: Arm 2

SUMMARY:
A study to assess the safety and efficacy of moxifloxacin compared to that of amoxicillin-clavulanic acid for the treatment of subjects with acute exacerbation of chronic bronchitis.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with chronic bronchitis
* Male or female subjects, >=60 years old
* Post bronchodilator forced expiratory volume in one second (FEV1) less than or equal to 60% predicted and FEV1 / forced vital capacity (FVC) less than 70% at enrollment
* Documented history of 2 or more AECB episodes, within 12 months of study enrollment, requiring a course of systemic antibiotics and/or systemic corticosteroids
* All symptoms/signs must be present and confirmed by the Investigator:

  * increase in dyspnea
  * purulent sputum
  * increase in sputum volume
* Current or past cigarette smoker with equal to or greater than 20 pack year smoking history
* Subjects must be exacerbation free for at least 30 days prior to enrollment
* Subjects must be willing and able to complete the questionnaires and subject booklet without assistance

Exclusion Criteria:

* Known hypersensitivity to quinolones, ß lactams, or to any of the excipients of the study drugs
* Known to have congenital or acquired QT prolongation
* Known to have clinically relevant bradycardia
* Known to have clinically relevant heart failure with reduced left ventricular ejection fraction
* Known to have previous history of symptomatic arrhythmias
* Taking QT prolonging drugs, for example Class Ia or III antiarrhythmic agents or other QT prolonging drugs
* Known electrolyte disturbances that are not controlled, particularly uncorrected hypokalemia
* Known history of hereditary problems of galactose intolerance, the Lapp lactase deficiency, or glucose galactose malabsorption
* History of a tendon disease/disorder
* Known history of liver dysfunction (Child-Pugh C), including known elevated transaminase levels (alanine aminotransferase [ALT] and/or aspartate aminotransferase [AST] >5 times the upper limit of normal [5 x ULN])
* Known severe renal impairment with glomerular filtration rate of <30 mL/min
* Known neutropenia (neutrophil count <1000/mm3) caused by immunosuppressive therapy or malignancy
* Known to have Acquired Immunodeficiency Syndrome (AIDS) (CD4 count of <200/mm3), or be human immunodeficiency virus (HIV) positive and receiving highly active anti retroviral therapy (HAART) (testing for HIV is not mandatory)
* Known chronic asthma (>15% reversibility or at least 200 mL), bronchial carcinoma, active pulmonary tuberculosis, known diffuse bronchiectasis, cystic fibrosis, or pneumonia (a chest x ray is not mandatory)
* Known history of chronic colonization of pathogenic organisms resistant to moxifloxacin and/or amoxicillin clavulanic acid (eg, P. aeruginosa, methicillin resistant Staphylococcus aureus)
* Receiving long term (>4 consecutive weeks) systemic corticosteroid treatment (>10 mg/day of prednisolone or equivalent)
* Received short course of systemic corticosteroid treatment within 30 days prior to enrollment
* Life expectancy of less than 6 months
* Receiving systemic antibacterial therapy within 30 days prior to study enrollment
* Requiring concomitant systemic antibacterial agents
* Requiring home ventilatory support (subjects requiring home/portable oxygen therapy or continuous positive airway pressure (CPAP) for sleep apnea are not excluded) and/or those who have a tracheotomy in situ
* History of liver function disorders following previous treatment with amoxicillin-clavulanic acid
* Receiving disulfiram therapy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1372 (Actual)
Dates: Start 2008-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Clinical failure at 8 weeks post therapy | At day 63

SECONDARY OUTCOMES:
Clinical failure rates | Through to day 35
Bacteriological eradication rates | Through to day 63
Clinical failure rates for subjects with positive sputum culture at enrollment | Through to day 63
Weekly mean symptom scores measured by the AECB SS | Through to day 63
Rates and speed of symptom relief measured by the AECB SS | Through to day 63
Clinical failure rates for subjects with co-administration of systemic corticosteroids (stratum 1) | Through to day 63
Clinical failure rates for subjects without co-administration of systemic corticosteroids (stratum 2) | Through to day 63
Need for any change in dosage or additional respiratory medication such as bronchodilators and inhaled steroids, excluding short acting bronchodilators | Through to day 63
Improvement in symptoms burden measured by the AECB SS | Through to day 63
Improvement in health related QoL measured by the SGRQ | Through to day 63
spirometry tests will be compared between treatment groups | Through to day 63
HCRU relat. to chronic bronchitis management incl. rescue med., concomitant med., therap. adjuncts, diagn. procedures, other medical care/medical staff requirement, hospitalizations (incl. ward and duration), and work productivity and activity impairment | Through to day 63
Safety and tolerability of moxifloxacin versus amoxicillin clavulanic acid, with particular attention to rates of diarrhea | Through to day 63

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (178):
- Les Escaldes, Andorra
- Argentina (5):
  - Quilmes, Buenos Aires
  - San Juan Bautista, Buenos Aires
  - Buenos Aires, Ciudad Auton. de Buenos Aires
  - San Miguel de Tucumán, Tucumán Province
  - Vicente López
- Australia (5):
  - Concord, New South Wales
  - Brisbane, Queensland
  - Adelaide, South Australia
  - Woodville, South Australia
  - Nedlands, Western Australia
- Belgium (8):
  - Aalst
  - Antwerp
  - Bruxelles - Brussel
  - Halen
  - Lommel
  - Moerkerke
  - Namur
  - Yvoir
- Brazil (3):
  - Juiz de Fora, Minas Gerais
  - Porto Alegre, Rio Grande do Sul
  - São Paulo, São Paulo
- Canada (15):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Kelowna, British Columbia
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Saint John, New Brunswick
  - Antigonish, Nova Scotia
  - Sydney Mines, Nova Scotia
  - Burlington, Ontario
  - Hamilton, Ontario
  - London, Ontario
  - Toronto, Ontario
  - Longueuil, Quebec
  - Montreal, Quebec
  - Sherbrooke, Quebec
- Chile (3):
  - Santiago
  - Valparaíso
  - Viña del Mar
- China (8):
  - Guangzhou, Guangdong
  - Changsha, Hunan
  - Shengyang, Liaoning
  - Shenyang, Liaoning
  - Chengdu, Sichuan
  - Beijing
  - Shanghai
  - Tianjin
- Colombia (5):
  - Cali, Cauca Department
  - Bogotá
  - Bucaramanga
  - Cali
  - Medellín
- Croatia (4):
  - Osijek
  - Petrinja
  - Rijeka
  - Zagreb
- Czechia (6):
  - Kyjov
  - Lovosice
  - Neratovice
  - Pardubice - Trnova
  - Praha - Malesice
  - Praha - Troja
- France (4):
  - Marseille
  - Mont-de-Marsan
  - Nice
  - Perpignan
- Germany (19):
  - Bad Dürrheim, Baden-Wurttemberg
  - Augsburg, Bavaria
  - Cottbus, Brandenburg
  - Rüdersdorf, Brandenburg
  - Zossen, Brandenburg
  - Hamburg, Hamburg
  - Frankfurt am Main, Hesse
  - Fulda, Hesse
  - Neubrandenburg, Mecklenburg-Vorpommern
  - Lüdenscheid, North Rhine-Westphalia
  - Neuwied, Rhineland-Palatinate
  - Böhlen, Saxony
  - Delitzsch, Saxony
  - Dresden, Saxony
  - Leipzig, Saxony
  - Meissen, Saxony
  - Bad Segeberg, Schleswig-Holstein
  - Lübeck, Schleswig-Holstein
  - Berlin, State of Berlin
- Greece (5):
  - Athens, Attica
  - Mezourlo, Larissa
  - Rio, Patras
  - Athens
  - Ioannina
- Hong Kong (2):
  - Hong Kong
  - Kowloon
- Indonesia (3):
  - Bandung
  - Jakarta
  - Surabaya
- Ireland (5):
  - Killarney, Kerry
  - Longford, Longford
  - Enniscorthy, Wexford
  - Gorey, Wexford
  - Bray, Wicklow
- Italy (8):
  - Pregiato Di Cava Dei Tirreni, Salerno
  - Busto Arsizio, Varese
  - Bussolengo, Verona
  - Ascoli Piceno
  - Catania
  - Chieti
  - Milan
  - Perugia
- Latvia (5):
  - Krāslava
  - Riga
  - Talsu
  - Valmiera
  - Ventspils
- Lithuania (4):
  - Kaunas
  - Klaipėda
  - Šiauliai
  - Vilnius
- Mexico (6):
  - Chihuahua City, Chihuahua
  - Guadalajara, Jalisco
  - Monterrey, Nuevo León
  - Huixquilucan, State of Mexico
  - Mérida, Yucatán
  - Zacatecas City, Zacatecas
- Netherlands (5):
  - Eindhoven, North Brabant
  - Heerlen
  - Hoofddorp
  - Meppel
  - Utrecht
- Pakistan (3):
  - Karachi, Sindh
  - Islamabad
  - Karachi
- Peru (3):
  - Lima, Lima Province
  - Callao
  - Lima
- Philippines (2):
  - Manila
  - Quezon City
- Portugal (8):
  - Coimbra, Coimbra District
  - Torres Vedras, Lisbon District
  - Matosinhos Municipality, Porto District
  - Vila Nova de Gaia, Porto District
  - Lisbon
  - Porto
  - S. Martinho Do Bispo
  - Santarém
- South Africa (12):
  - Port Elizabeth, Eastern Cape
  - Bloemfontein, Freestate
  - Benoni, Gauteng
  - Centurion, Gauteng
  - Kempton Park, Gauteng
  - Pretoria, Gauteng
  - Durban, KwaZulu-Natal
  - Thabazimbi, Limpopo
  - Witbank, Mpumalanga
  - Cape Town, Western Cape
  - Paarl, Western Cape
  - Somerset West, Western Cape
- Spain (7):
  - Badalona, Barcelona
  - Barcelona, Barcelona
  - Sant Boi de Llobregat, Barcelona
  - Guadalajara, Guadalajara
  - Palma de Mallorca, Illes Baleares
  - Madrid, Madrid
  - Requena, Valencia
- Switzerland (9):
  - Laufen, Basel-Landschaft
  - Oberwil, Basel-Landschaft
  - Aarau, Canton of Aargau
  - Binningen, Canton of Basel-City
  - Bern, Canton of Bern
  - Zurich, Canton of Zurich
  - Basel
  - Thun
  - Wettingen
- Thailand (3):
  - Chiang Mai, Thailand
  - Bangkok
  - Nonthaburi
- United Kingdom (2):
  - Glasgow, Stratchclyde
  - Coventry, Warwickshire

REFERENCES:
- [Result] Wilson R, Anzueto A, Miravitlles M, Arvis P, Farago G, Haverstock D, Trajanovic M, Sethi S. A novel study design for antibiotic trials in acute exacerbations of COPD: MAESTRAL methodology. Int J Chron Obstruct Pulmon Dis. 2011;6:373-83. doi: 10.2147/COPD.S21071. Epub 2011 Jun 29. PMID 21760724
- [Derived] Wilson R, Anzueto A, Miravitlles M, Arvis P, Haverstock D, Trajanovic M, Sethi S. Prognostic factors for clinical failure of exacerbations in elderly outpatients with moderate-to-severe COPD. Int J Chron Obstruct Pulmon Dis. 2015 Jun 2;10:985-93. doi: 10.2147/COPD.S80926. eCollection 2015. PMID 26082623
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/